CLINICAL TRIAL: NCT05146765
Title: Efficacy of a Digital Therapeutic for People With Dysarthria After Stroke; Pilot Trial
Brief Title: Efficacy of a Digital Therapeutic for People With Dysarthria After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ewha Womans University Seoul Hospital (Other)
Responsible Party: Principal Investigator, Tae-Jin Song, MD, PhD, Principal investigator, Department of neurology, Seoul Hospital, Ewha Womans University College of Medicine, Ewha Womans University Seoul Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D-ST01
Record Dates: First submitted 2021-11-14; First posted 2021-12-07 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Dysarthria as Late Effect of Stroke
Keywords: Dysarthria; Stroke; digital therapeutics; Speech Disorders; Language Disorders; speech rehabilitation; application; Post-stroke dysarthria
MeSH Terms: conditions — Dysarthria; Stroke; Speech Disorders; Language Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Pilot trial
Who Masked: Participant
Masking Description: Outcome Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive treatment as usual along with the speech therapy app.
  Interventions: Device: Mobile application; Other: Treatment as usual
- Control (No Intervention): The control group will receive treatment as usual only.

INTERVENTIONS:
Device: Mobile application — Device: Use of mobile application Participants will be instructed to use the speech therapy app for 30 minutes to one hour per day over a 4-week period.
  Arms: Intervention
Other: Treatment as usual — The patients will follow the treatment as usual, including conventional stroke therapy if needed based on the medical guidelines.
  Arms: Intervention

SUMMARY:
This pilot trial will establish the feasibility of a new digitized speech rehabilitation developed for patients with post-stroke dysarthria. For this study, participants will be instructed to use the speech therapy app for 30 minutes to 1 hour per day over a 4-week period.

DETAILED DESCRIPTION:
A total of 40 patients with post-stroke dysarthria will be recruited and randomly divided into intervention and control groups.

Patients in the intervention group will be instructed to receive speech treatments including oro-motor exercise, phonation, articulation, resonance, syllable repetition, and reading exercise (App on mobile devices). Daily sessions will be provided during a 4-week period. Both groups will also receive treatment as usual. The aim of the study is to investigate the efficacy of mobile-based speech therapy in patients with dysarthria in the acute phase following stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Neurologically stable, as determined by the clinician.
2. Onset of stroke within four weeks prior to randomization.
3. Diagnosis of dysarthria caused by stroke as confirmed by a stroke specialty neurologist.
4. Maintains enough cognitive function to use the speech therapy application without problems, as determined by a Mini-Mental State Exam score of 26 ≥ within 1 month prior to randomization.
5. Capable of walking or moving alone or with the assistance of a walking aid (e.g., walkers, canes, or wheelchairs).
6. Must have intact vision, hearing, communication skills, and motor skills, as well as comprehension sufficient to proceed with assessment, as judged by the clinician.

Exclusion Criteria:

1. Unable to measure articulatory or orofacial functions due to organic causes/lesions in articulatory and cervical structure.
2. Has comorbid neurological conditions that, in the opinion of the investigator, could impair study participation, such as dementia (Alzheimer's disease, vascular dementia, Central Nervous System Infection [e.g., Human Immunodeficiency Virus, syphilis], Creutzfeld-Jacob disease, etc.), Pick's disease, Huntington's disease, or Parkinson's disease.
3. Has a Mini-Mental State Exam score of 26 or below at the time of screening.
4. Has a Clinical Dementia Rating score of 1 ≥ or a Global Deterioration Scale score of 3 ≥ at the time of screening.
5. Received dementia treatment within 3 months of screening.
6. Takes medication that may impact cognitive function during the clinical trial period.
7. Co-medication is prohibited during the entire trial period for the following medications: drugs for dementia treatment, Central Nervous System stimulants, anticholinergics, tricyclic antidepressants, typical antipsychotics, and sleeping pills (excluding rapid-acting sleeping pills).
8. Co-medication is permitted if continued use of the following medications has been at a stable dose for 2 months prior to randomization: atypical antipsychotics, anxiolytics, antidepressants (excluding tricyclic antidepressants), thyroid hormone, and rapid-acting sleeping pills.
9. Is uneducated or illiterate.
10. Has been diagnosed with a serious mental illness such as severe depression, schizophrenia, alcohol addiction, or drug addiction.
11. Unable to use D-ST01 due to severe speech impairment, as determined by the clinician.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Speech intelligibility | Baseline, 4weeks
  Speech intelligibility is evaluated with a score of 0 (normal), 1 (intelligible, some differences noticeable), 2 (intelligible, noticeably different), 3 (intelligible with careful listening, some unintelligible), 4 (difficult to understand, many words unintelligible), 5 (usually unintelligible), or 6 (unintelligible).

SECONDARY OUTCOMES:
The percent change in score on the Urimal Test of Articulation and Phonology 2 (UTAP2) | Baseline, 4weeks
  he UTAP2, an essential tool for determining articulatory proficiency, will be employed to evaluate the Percentage of Consonants Correct (PCC), a crucial metric for identifying irregularities in articulation. Study participants will be instructed to read all 30 words from the UTAP2 word-level test. Following this, evaluators will calculate the PCC, expressed as a percentage, using the 94 consonants included in these words. This methodology acknowledges that a PCC of 0% signifies lower articulatory accuracy, whereas a PCC of 100% reflects a higher level of precision.

OTHER OUTCOMES:
National Institute of Health Stroke Scale (NIHSS) | Baseline, 4weeks
  NIHSS will be used to assess stroke-related neurologic deficits. The NIHSS scale is made up of 11 different elements that evaluate specific abilities; level of consciousness (LOC), best gaze, visual field, facial palsy, motor arm, motor leg, limb ataxia, sensory, best language, dysarthria, extinction, inattention. The score ranges from 0 to 42; higher scores indicate more severe stroke symptoms.
Patient Health Questionnaire-9 (PHQ-9) | Baseline, 4weeks
  The PHQ-9 is a nine-item self-reported questionnaire that is used to assess depressive symptoms. The score ranges from 0 to 27, with lower scores indicating less depressive severity.
Generalized Anxiety disorder-7 | Baseline, 4weeks
  GAD-7(Generalized Anxiety disorder-7) will be used to assess anxiety. The GAD-7(Generalized Anxiety disorder-7) is a seven-item self-reported questionnaire that evaluates anxiety symptoms. The score ranges from 0 to 21, with lower scores indicating lower anxiety symptoms.
Euro Quality of Life (EQ-5D) | Baseline, 4weeks
  EQ-5D will be used to assess the quality of life. The EQ-5D is a self-report questionnaire that measures health-related quality of life. The questionnaire consists of five dimensions: mobility, self-care, ordinary activities, discomfort, and mood state related to anxiety or depression. The responses indicate three levels of severity ("no problems", "some problems", and "extreme problems") within each EQ-5D dimension.
Modified Computer Self-Efficacy Scale (mCSES) | Baseline, 4weeks
  mCSES will be used to assess participants' perceptions of self-efficacy with respect to using a computerized system. The mCSES is a 10-item self-reported questionnaire. The score ranges from 0 to 100; higher scores indicate a stronger sense of personal competence.

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Jin Song, MD, PhD, Principal Investigator — Department of Neurology, Ewha University College of Medicine, Seoul, Republic of Korea
Locations (1):
- Ewha Womans University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim Y, Kim M, Kim J, Song TJ. Smartphone-Based Speech Therapy for Poststroke Dysarthria: Pilot Randomized Controlled Trial Evaluating Efficacy and Feasibility. J Med Internet Res. 2024 Apr 25;26:e56417. doi: 10.2196/56417. PMID 38509662